CLINICAL TRIAL: NCT07034742
Title: Exploratory Study on the Application of Molecular Residual Disease (MRD) in Postoperative Treatment of Gastric Cancer
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Dong Bing Zhao, MD, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25/099-5045
Record Dates: First submitted 2025-06-14; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Gastric Adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GC patients (Experimental)
  Interventions: Drug: Intraperitoneal chemotherapy PLUS systemic chemotherapy

INTERVENTIONS:
Drug: Intraperitoneal chemotherapy PLUS systemic chemotherapy — Intraperitoneal chemotherapy (fluorouracil + nab-paclitaxel + cisplatin + interleukin-2) PLUS systemic chemotherapy (SOX regimen: oxaliplatin + tegafur-gimeracil-oteracil potassium)

SUMMARY:
Gastric cancer is one of the most prevalent and lethal malignancies in China. The majority of patients are diagnosed at the locally advanced stage. Despite standard treatment involving radical resection combined with adjuvant chemotherapy, approximately 40% of patients experience recurrence and metastasis, with peritoneal metastasis accounting for nearly half of these cases.

Building upon our team's previous establishment of next-generation sequencing (NGS) technology for detecting molecular residual disease (MRD) in peritoneal lavage fluid and blood, this project aims to guide systemic chemotherapy with or without intraperitoneal chemotherapy for locally advanced gastric cancer patients based on the results of peritoneal lavage fluid MRD testing. We will investigate whether intraperitoneal chemotherapy can reduce the peritoneal metastasis rate in patients testing positive for MRD in peritoneal lavage fluid. The ultimate goal is to propose a novel diagnostic and therapeutic strategy for post-operative adjuvant treatment of gastric cancer, addressing this critical clinical challenge.

Patients testing negative for MRD in peritoneal lavage fluid will be enrolled in an observational cohort study. This cohort will explore the concordance between blood-based MRD positivity and actual clinical recurrence and metastasis. The objectives are to determine whether blood-based MRD can predict the occurrence of non-peritoneal metastasis after surgery and whether it can be used to evaluate the efficacy of post-operative systemic chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma, mucinous adenocarcinoma, or signet ring cell carcinoma of the stomach or gastroesophageal junction (GEJ).
* Clinical stage cT4NanyM0, deemed suitable for radical resection.
* Age between 18 and 75 years.
* ECOG performance status of 0 or 1.
* No prior neoadjuvant therapy and strong patient/family preference for primary surgery.
* Adequate organ function defined as:

Absolute neutrophil count (ANC) > 1.5 x 10⁹/L (or > 1500/µL)；Hemoglobin (Hb) > 90 g/L；Platelet count (PLT) > 100 x 10⁹/L (or > 100,000/µL)；Alanine aminotransferase (ALT) and Aspartate aminotransferase (AST) < 2.5 x Upper Limit of Normal (ULN)；Total bilirubin (TBIL) < 1.5 x ULN；Serum creatinine (Cr) < 1.0 x ULN

* Good compliance and willingness to undergo long-term follow-up.
* Provision of signed written informed consent.

Exclusion Criteria:

* Pathological specimens containing >10% of other histological components (e.g., squamous cell carcinoma, neuroendocrine carcinoma, etc.).
* Uncontrolled gastrointestinal obstruction or recurrent bleeding.
* Inability to swallow oral medications.
* Active infection requiring systemic therapy.
* Moderate to severe cirrhosis due to any cause.
* Cardiac function classified as NYHA class > I.
* History of myocardial infarction, unstable angina, stroke, or uncontrolled arrhythmia.
* Anticipated inability to tolerate postoperative adjuvant chemotherapy.
* Concurrent medical conditions that contraindicate chemotherapy.
* Pregnancy or lactation; history of psychiatric illness; poor compliance.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
2-year peritoneal metastasis-free survival rate | 2-year

CONTACTS AND LOCATIONS:
Locations (1):
- Chaoyang District, Panjiayuan Nanli NO.17, Beijing, China

IPD SHARING:
Plan to Share IPD: No